CLINICAL TRIAL: NCT06307964
Title: Intra-Hepatic Microbiota in Alcoholic Hepatitis
Acronym: HepMAH
Status: Recruiting | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL23_1137; ID-RCB (Other: 2024-A00480-47)
Record Dates: First submitted 2024-03-06; First posted 2024-03-13 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-01

CONDITIONS: Cirrhosis; Alcoholic Liver Disease; Alcoholic Hepatitis
Keywords: alcoholic hepatis; bacterial translocation; microbiota; 16S rRNA; intra-hepatic microbiota; cirrhosis; alcoholic liver disease
MeSH Terms: conditions — Fibrosis; Liver Diseases, Alcoholic; Hepatitis, Alcoholic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Three types of biospecimen would be obtained:
  * A fragment of the diagnostic transjugular liver biopsy (D0)
  * Plasma samples at D0, and at 1 and 6 months after liver biopsy if possible
  * Fecal samples at D0, and at 1 and 6 months after liver biopsy if possible
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Alcoholic hepatitis: Patients with histologically proven AH (after transjugular liver biopsy procedure and histological assessment).
  Interventions: Procedure: Biological sampling
- No alcoholic hepatitis: Patients with initially suspected AH (excessive alcohol consumption and modified Maddrey score > 32) but no AH at the histological evaluation of liver biopsy.
  It corresponds to patients with decompensated alcoholic liver disease but no AH.
  Interventions: Procedure: Biological sampling

INTERVENTIONS:
Procedure: Biological sampling — * A fragment of the diagnostic transjugular liver biopsy (D0)
  * Plasma samples at D0, and at 1 and 6 months after liver biopsy if possible
  * Fecal samples at D0, and at 1 and 6 months after liver biopsy if possible

SUMMARY:
Alcoholic hepatitis (AH) is a serious complication of alcoholic liver disease (ALD). The histological presentation of AH is characterized by neutrophilic lobular inflammation, macrovesicular steatosis, hepatocyte ballooning and necrosis and the presence of Mallory bodies. In cases of severe HA, defined by a modified Maddrey score of 32 or above, mortality at 1 month is estimated at between 10 and 50%. The only treatment to reduce early mortality is corticosteroid therapy. However, only 60% of patients respond to corticosteroids, and no benefit has been demonstrated on late mortality. Identifying new therapeutic targets is therefore a major challenge in this disease.

Numerous pre-clinical studies and human data suggest the involvement of the intestinal microbiota in the pathogenesis of AH. Translocation of viable bacteria and microbial products from the digestive tract to the liver contributes to local and systemic inflammation, hepatocyte death and fibrogenesis. However, the intrahepatic microbial environment has never been characterized in HA.

The study hypothesis is that the intrahepatic microbiota is modulated by bacterial translocation and is associated with clinical outcomes.

The aim of this study is to determine the composition of the intrahepatic (obtained from transjugular liver biopsy), blood and fecal microbiota in patients with suspected severe AH from a monocentric prospective cohort in the Hepatology Department at Croix-Rousse Hospital (Lyon). Fifty consecutive patients with clinical suspicion of AH and indication for transjugular liver biopsy will be included. About thirty-five patients are expected in the confirmed AH group, and 15 in the group "alcoholic liver disease with no AH", based on data from the literature. The composition of the various microbiota will be determined by sequencing the 16S rRNA gene, and the results will be correlated with clinical data (corticosteroid sensitivity, overall survival, transplant-free survival, MELD score in particular) and histological data.

This exploratory study will enable to analyze the intra-hepatic microbiota, and to study its link with intra-hepatic inflammation and the clinical course of patients with AH. The data generated by HepMAH will thus help identify potential new therapeutic targets linked to the gut microbiota, and provide a scientific basis for the development of therapeutic interventions targeting the microbiota in HA.

ELIGIBILITY:
Inclusion Criteria:

* Patients suffering from alcoholic liver disease and clinical suspicion of alcoholic hepatitis (subacute jaundice, heavy alcohol consumption active or weaned for ≤ 3 months, modified Maddrey score ≥32) and indication for diagnostic transjugular liver biopsy;
* Non-objection obtained from the patient or trusted person in case of impaired judgment or consciousness before performing liver biopsy;
* Aged ≥ 18 years at the time of study entry;

Exclusion Criteria:

* Patients who were treated with antibiotics or probiotics between the 15th day and 72 hours prior to liver biopsy, with the exception of antibiotics used for the prophylaxis of ascites infection or hepatic encephalopathy
* Contraindication to transjugular liver biopsy (hepatocellular carcinoma on predicted puncture site)
* Pregnant, parturient or breast-feeding women
* Persons deprived of their liberty by judicial or administrative decision
* Adults under legal protection (guardianship, curators)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A prospective observational multicentric cohort will be conducted at Croix Rousse Hospital (Lyon, France), in the Hepatology and Intensive Care Units.
  Fifty consecutive patients hospitalized in either of these units for clinical suspicion of alcoholic hepatitis and indication for transjugular liver biopsy will be included.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-07-23 (Actual); Primary Completion 2028-01-23 (Estimated); Study Completion 2028-07-23 (Estimated)

PRIMARY OUTCOMES:
Microbiota composition | At Day 0, 1 month and 6 months
  Intrahepatic, blood and fecal microbiota composition will be assessed by 16S rRNA sequencing (MiSeq Illumina). Microbiota analysis will be performed on the fragment of transjugular liver biopsy collected for the purpose of the study, and on plasma and fecal samples after bacterial DNA extraction.
  Bioinformatics analysis will be carried out using Qiime2, LeFSE (Conda) and the Maaslin2 package (v3.16; R software). Microbiota profiles determined at the genus taxonomic level will be compared between the two groups (proven AH and no AH).

CONTACTS AND LOCATIONS:
Overall Officials: François VILLERET, M.D., Ph.D., Study Chair — Hospices Civils de Lyon, Croix Rousse Hospital, Hepatology department
Locations (1):
- Hospices Civils de Lyon, Croix Rousse Hospital, Lyon, France